CLINICAL TRIAL: NCT02413814
Title: Computerized Anger-Reduction Treatment for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34DA035944-01A1 (NIH)
Record Dates: First submitted 2015-03-09; First posted 2015-04-10 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Anger; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anger Reduction Treatment (Experimental): The treatment consists of eight 30-minute IBM sessions. Participants will be presented with ambiguous scenarios and asked imagine themselves in these situations. In the first task, the scenario will be followed by a benign interpretation of the situation. Participants will answer a comprehension question designed to have participants endorse this benign interpretation. In the second task, participants will be presented with a word denoting an interpretation with either a negative/hostile or positive/benign connotation. Following this word, an ambiguous scenario will appear. Participants will indicate whether the word and the scenario were related. They will receive feedback training them to endorse positive interpretations and reject negative interpretations.
  Interventions: Behavioral: Anger Reduction Treatment
- Control Condition (Placebo Comparator): Participants assigned to the control condition will complete eight computerized sessions consisting of psychoeducation on healthy behaviors (i.e., topics of exercise, diet, hygiene, social support, healthy activities, and sleep, taken from protocols developed from our ongoing research). These participants will also view relaxing videos consisting of brief guided meditation instructions, pictures of nature scenes, and soft music. These sessions (psychoeducation and relaxing videos) will be matched for time with the active treatment condition, lasting 30 minutes each.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Anger Reduction Treatment — Eight 30-minute sessions of interpretation modification to reduce angry interpretation biases.
  Arms: Anger Reduction Treatment
Behavioral: Control Condition — Eight 30-minute sessions of informative videos on healthy living and relaxation videos.
  Arms: Control Condition

SUMMARY:
Problematic anger is a strong predictor of failed attempts at smoking cessation. The investigators proposed study seeks to evaluate whether a novel 8-session computerized anger-reduction treatment improves quit rates among smokers. Smokers with elevated trait anger will be administered transdermal nicotine patch therapy and either anger-reduction treatment or a control intervention. They will be assessed throughout treatment and up until three months after a scheduled mid- treatment quit date. The investigators propose to test whether, compared to the control condition, the anger-reduction treatment will lead to: 1) greater reductions in anger and 2) greater abstinence rates at post-cessation and at follow-up assessments. The investigators will also test whether changes in anger-related symptoms account for group differences in abstinence rates.

DETAILED DESCRIPTION:
The current proposal seeks to evaluate an eight-session, computerized, anger-focused intervention for smokers (Anger Reduction Treatment or ART). The investigators will administer this intervention to smokers (N = 114) who are interested in quitting and have elevated levels of trait anger. Participants will be randomly assigned to receive either: (1) computerized ART, consisting of interpretation bias modification, or (2) a computerized control condition, which consists of health education and relaxing video clips. The computerized sessions (eight total) will take place twice a week for four weeks. All participants will have a scheduled quit date for the beginning of the third week of treatment (i.e., at mid-treatment). All participants will also receive nicotine patch therapy to use at their scheduled quit date. Anger symptoms, smoking cravings, and smoking frequency will be assessed throughout treatment. Smoking status, anger, and other measures of negative affect will also be assessed at baseline and regularly for 12-weeks following the scheduled quit date.

The investigators will test whether, compared to the control condition, the anger-reduction treatment will lead to: 1) greater reductions in anger and 2) greater abstinence rates at post-cessation and at follow-up assessments. The investigators will also test whether changes in anger-related symptoms account for group differences in abstinence rates.

ELIGIBILITY:
Inclusion Criteria:

* Elevated levels of trait anger (scoring 22 or higher on the STAXI-trait)
* Currently smoking an average of 8 cigarettes per day
* Must be a regular (daily) smoker for at least 1 year
* Willing to make a serious attempt to quit smoking
* Must report motivation to quit in the next month (30 days) of at least 5 on a 10 point scale (0 = no motivation and 10 = extreme motivation)
* Have not decreased the number of cigarettes by more than half in the past six months
* Must be an English speaker

Exclusion Criteria:

* Current substance dependence (excluding nicotine dependence)
* Current use of other tobacco products
* Currently receiving cognitive therapy or therapy for problematic anger
* Evidence of serious suicidal intent requiring hospitalization or immediate treatment
* Limited mental competency and the inability to give informed, written consent
* Evidence of psychotic-spectrum disorders
* Changes in medication over the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
State-Trait Anger Expression Inventory-2 (STAXI-2; Spielberger, 1999) state and trait subscales | up to 14-weeks following treatment initiation.
Self-reported smoking frequency | up to 14-weeks following treatment initiation.
Carbon monoxide levels | up to 14-weeks following treatment initiation.

SECONDARY OUTCOMES:
Minnesota Nicotine Withdrawal Scale (Hughes & Hatsukami, 1986) | up to 14-weeks following treatment initiation.
Beck Depression Inventory-II (Beck, Steer, & Brown, 1996) | Baseline and regularly for 14-weeks following treatment initiation.
Clinical Anger Scale (CAS; Snell, Gum, Shuck, Mosley, & Hite, 1995) | up to 14-weeks following treatment initiation.
WSAP-Hostility Scale (Dillon, Cougle, & Fincham, 2015) | up to 14-weeks following treatment initiation.
Hostile Automatic Thoughts Scale (Snyder, Crowson, Houston, Kurylo, & Piorier, 1997) | up to 14-weeks following treatment initiation
Questionnaire of Smoking Urges (Tiffany & Drobes, 1991) | up to 14-weeks following treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse R Cougle, Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State University, Department of Psychology, Tallahassee, Florida, United States